CLINICAL TRIAL: NCT01522586
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dosing, Dose-escalation Clinical Phase 1 Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of DWP09031
Brief Title: Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of DWP09031
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: change development strategy
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: DWP09031
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DWP09031 (Experimental): DWP09031 50mg/100mg/400mg/200mg/800mg/1200mg/1600mg/2000mg single dosing
  Interventions: Drug: DWP09031
- Placebo (Placebo Comparator): placebo comparator 50mg/100mg/400mg/200mg/800mg/1200mg/1600mg/2000mg single dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP09031 — DWP09031 50mg/100mg/400mg/200mg/800mg/1200mg/1600mg/2000mg single dosing
  Arms: DWP09031
Drug: Placebo — placebo comparator 50mg/100mg/400mg/200mg/800mg/1200mg/1600mg/2000mg single dosing
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of orally administrated DWP09031 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects aged 20 to 45 years
2. The subject has Broca's index ≤ 20%
3. A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)
4. A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints

Exclusion Criteria:

1. A subject with sign or symptoms or previously diagnosed disease of liver (viral hepatitis), digestive system, cardiovascular, kidney, respiratory, endocrinology, neurology, immune system, hematology, and psychology function or other significant diseases and history or suspicion of current drug abuse and alcohol abuse
2. A subject who shows vital signs with the number of systolic blood pressure of ≥141 mmHg or ≤89 mmHg, and the number of diastolic blood pressure of ≥91mmHg
3. A subject who shows the following result in clinical laboratory test:

   AST,ALT>1.25 times of the upper limit of normal range PR ≥ 210 msec QRS ≥ 120 msec QT ≥ 500 msec QTcF ≥ 450 msec creatinine clearance ≤ 80mL/min
4. Subject who has taken other clinical or licensed medication from another clinical trial within an 90-day period prior to the first administration of the study medication (The last administration of the medication is considered as an end point of the previous clinical trial).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety&tolerability | -1d, 0 (predose), 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h, 8d (post-study visit)
  Adverse events, Physical exam, Vital sign, laboratory(CBC,chemistry,U/A etc)

SECONDARY OUTCOMES:
Pharmacokinetics | 0 (predose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 ,24 ,36, 48 h
  Cmax, AUClast, AUCinf, t1/2, CL/F, Vd/F

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, Professor, Principal Investigator — BUSAN PAIK HOSPITAL
Locations (1):
- Inje University College of Medicine Busan Paik Hospital, Busan, Busanjin-gu, South Korea